CLINICAL TRIAL: NCT05175404
Title: Use of 18F-PSMA-11 PET for Detection of Lesions in Iodine Refractory Thyroid Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-09501
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-11

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overal Trial (Other): only one arm in this trial
  Interventions: Diagnostic Test: PET/CT scan F18-PSMA-11

INTERVENTIONS:
Diagnostic Test: PET/CT scan F18-PSMA-11 — PET/CT scan with F18-PSMA-11

SUMMARY:
Determine the diagnostic value of 18F-PSMA-11 in patients with iodine refractory thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older.
* Signed Informed Consent.
* Subject is diagnosed with a histologically confirmed differentiated thyroid carcinoma, that is considered RAI refractory. There is evidence of persisting or recurrent disease, based on serum thyroglobulin levels and/or medical imaging.
* Subject should have a routine clinical 18F-FDG PET/CT performed within two months prior to the study scan.
* Female patients should be either post-menopausal, surgically sterile, or using highly effective contraceptives (methods that can achieve a failure rate of less than 1%: combined hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence).

Exclusion Criteria:

* Patient has a known other active malignancy.
* Subject is potentially pregnant (urinary test can be performed in case of doubt) or breastfeeding.
* Patient is mentally or legally incapacitated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Demonstrate uptake of 18F-PSMA-11 in RAI-RTC | 60 minutes +- 5 minutes after injection 18F-PSMA-11
  Confirmation in PET-scan that lesions in RAI-RTC show uptake of 18F-PSMA-11, above background activity in the bloodpool.

SECONDARY OUTCOMES:
Perform a semi-quantitative analysis of radiotracer uptake in lesions. | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Perform a lesion detection rate analysis on organ level. | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Compare uptake of 18F-PSMA-11 in these patients to the uptake of 18F-FDG, on a lesion basis. | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Evaluate the sufficiency of uptake of 18F-PSMA-11 to consider therapy with 177Lu-PSMA in a subset of patients | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Compare the histological expression of PSMA on already available tumor samples with the uptake of lesions on PSMA PET. | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Analyse the correlation between the serum level of PSMA and the uptake on PSMA PET | 60 minutes +- 5 minutes after injection 18F-PSMA-11
Compare the histological expression of PSMA on already available tumor samples with the serum level of PSMA. | Within 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Ghent, Ghent, Belgium

REFERENCES:
- [Result] Van den Broeck B, Debacker JM, Bauters W, Creytens D, Ferdinande L, Huvenne W, Lapauw B, Schelfhout V, Van Laeken N, Verroken C. Potential application of [18F]AlF-PSMA-11 PET/CT in radioiodine refractory thyroid carcinoma. EJNMMI Res. 2024 Sep 12;14(1):82. doi: 10.1186/s13550-024-01148-9. PMID 39264376